CLINICAL TRIAL: NCT01322776
Title: Phase 1 and 2 Study of Combination Treatment of Bortezomib, Fludarabine and Cyclophosphamide in Patients With Recurrent Mantle Cell Lymphoma
Brief Title: Combination of Bortezomib, Fludarabine and Cyclophosphamide Treat Recurrent Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other); Zhejiang University (Other); West China Hospital (Other); Ruijin Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Peking University Cancer Hospital & Institute (Other); Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Huiqiang Huang, Sun Yat-sen University Cancer Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vel-FC-4003
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Mantle Cell Lymphoma Recurrent
Keywords: Mantle Cell Lymphoma; Recurrent; Bortezomib; Combination Treatment
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib,Fludarabine,Cyclophosphamide (Experimental)
  Interventions: Drug: Combination of Bortezomib, Fludarabine and Cyclophosphamide

INTERVENTIONS:
Drug: Combination of Bortezomib, Fludarabine and Cyclophosphamide — bortezomib 1.3mg/m^2 i.v. on days 1, 4, 8 and 11 of each 28-day cycle fludarabine 25mg/m^2 i.v. on days 1~3 of each 28-day cycle cyclophosphamide i.v. on days 1~2 of each 28-day cycle

SUMMARY:
This is a multi-center, single arm, open-label, prospective IIS study, which will enroll 40 recurrent MCL patients.The aim is to evaluate the efficacy and safety of bortezomib, fludarabine and cyclophosphamide treatment and also analyze the relationship between NF-kB activity and efficacy of bortezomib treatment and whether NF-kB activity can predict MCL progression.

DETAILED DESCRIPTION:
This is a multi-center, single arm, open-label, prospective IIS study, which will enroll 40 recurrent MCL patients.The aim is to evaluate the efficacy and safety of bortezomib, fludarabine and cyclophosphamide treatment and also analyze the relationship between NF-kB activity and efficacy of bortezomib treatment and whether NF-kB activity can predict MCL progression.

This study consists of three phases: screening/baseline phase, treatment phase and follow-up phase after the end of treatment.

At screening/baseline phase, investigators obtain informed consent form, check the inclusion/exclusion criteria and then collect the following data: demographics, medical history data, vital signs, ECG, MRI/CT/B-ultrasound/X-ray examinations, physical examination, laboratory examinations, pregnancy test (only female) and bone marrow biopsy and aspiration. Pathological diagnosis of mantle cell lymphoma should be established by lymph node biopsy or other tumor histopathological examination and immunophenotyping. At the same time, ECOG-performance status, Fact/GOG-Ntx questionnaire and NF-κB activity will be assessed.

During treatment period, patients will be treated with bortezomib, fludarabine and cyclophosphamide in a 28-day cycle. Patients achieve complete response (CR) or partial response (PR) can receive up to six cycles of VF (C) treatment, while those continue stable disease (SD) will be stopped after 4-cycle treatment and those with progressive disease (PD) will also be stopped after 2-cycle treatment. Due to adverse events, patients may receive reductions or deviate from the intended dose and duration of VF (C) treatment. These adjustments must be in accordance with the regulations in the protocol about the dose and time adjustment.

Maximum tolerated dose (MTD) of cyclophosphamide will be determined in accordance with the standard "3+3" method, testing three dose levels, 150mg/m2, 200mg/m2 and 250mg/m2. Cyclophosphamide dose escalation test will be conducted in the first cycle, with every three patients in a group. Patients' enrollment will be competed among different sites, but further step should be taken only after the 3 patients in one group complete the first cycle, their efficacy and safety have been completely evaluated, and the notification of going to next step by a CRO company. Subjects involved in the cyclophosphamide dose escalation test will continue initial cyclophosphamide dose during the entire study, except for possible dose adjustment determined by investigators due to DLT. After ascertaining MTD, new patients will be administrated with cyclophosphamide at the MTD. According to the dose escalation diagram, up to 18 patients will be involved in dose escalation phase. Subjects who discontinue the treatment due to causes other than DLT in the first cycle should be replaced by new participants to enter dose escalation test. DLT is defined as: a grade 4 neutropenia lasting longer than 7 days, a grade 4 thrombocytopenia, a neutropenic fever, or a grade 3 or above non-hematological toxicity (except for nausea, vomiting and alopecia); a grade 3 or above nausea, vomiting or diarrhea is considered as DLT only if still observed after treatment. Please refer to dose escalation diagram to conduct dose escalation trial.

Subjects will be followed up for 24 weeks after the end of chemotherapy. In this study, the primary efficacy endpoints are maximum tolerated dose (MTD) of cyclophosphamide in combination treatment with bortezomib and fludarabine, complete response rate (CR + CRu), overall response rate (ORR). Main indicators will be evaluated every 2 cycles in the treatment period and every 12 weeks in follow-up period.

Concomitant medications within 2 week before enrollment and during the study process need to be documented. All adverse events will be reported from the time a signed and dated informed consent form is obtained until 30 days following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older;
* Histologically confirmed MCL (Initial diagnosis in hospitals other than sites must be reconfirmed;
* Recurrent patients after first-line or second-line chemotherapy;
* At least including the following characteristic immunophenotype confirmed by immunohistochemistry: CD 20+, CD5+ and cyclin D1+;
* At least 1 measurable site of tumor（long diameter > 2.0 cm by physical examination or > 1.5cm on CT;
* No involvement of central nervous system;
* ECOG performance status ≤ 2，life expectancy>6 months;
* Within 14 days before enrollment，WBC > 3×10^9/L，neutrophils > 1.5×10^9/L，platelets > 75×10^9/L;
* ALT ≤ 2 × upper limit of normal (ULN)，AST ≤ 2×ULN，total bilirubin ≤ 2×ULN，serum creatinine ≤ 1.5×ULN，calculated creatinine clearance > 50ml/min;
* Female patients must be post menopausal, surgically sterile, or practicing an effective method of birth control;
* Male patients must agree to use an acceptable method of contraception for the duration of the study;
* All patients must have signed an informed consent document indicating that they understand the purpose and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Peripheral neuropathy or neuropathic pain of grade 2 or worse according to CTC AE 3.0;
* Prior treatment with bortezomib;
* Diagnosed as a malignancy other than MCL（Patients with completely resected basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy are not excluded;
* Any experimental or anti-cancer therapy within 4 weeks before the first dose of study drug (including rituximab, alemtuzumab or unconjugated therapeutic antibodies, radiation therapy, etc.);
* Fludarabine resistance or intolerance，exposure to fludarabine within 6 months before screening；History of allergic reaction to compounds containing boron, mannitol, fludarabine or cyclophosphamide;
* Patients with known diagnosis of active systemic infection, HIV or active hepatitis B (carriers of hepatitis B are permitted to enter study);
* Serious medical (e.g., cardiac failure [New York Heart Association: NYHA Class III or IV, or left ventricular ejection fraction: LVEF < 50%], active peptic ulceration, or uncontrolled diabetes mellitus) or psychiatric illness likely to interfere with participation in this clinical study;
* Pregnancy or lactation;
* Female or male patients of child-bearing potential who will not use adequate contraception during the course of the study;
* Other condition likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy will be assessed according to the CT scan and bone marrow aspirate and biopsy | 2cycle,28-day/cycle
  The International Working Group (IWG) published the guidelines for response criteria for lymphoma in 1999. These response criteria are based on the reduction in the size of the enlarged lymph node as measured by CT scan and the extent of bone marrow involvement that is determined by bone marrow aspirate and biopsy.

SECONDARY OUTCOMES:
Maximum Tolerated Dose（MTD）of Cyclophosphamide | 6 months
  Maximum tolerated dose (MTD) of cyclophosphamide will be determined in accordance with the standard "3+3" method, testing three dose levels, 150mg/m^2, 200mg/m^2 and 250mg/m^2. Cyclophosphamide dose escalation test will be conducted in the first cycle, with every three patients in a group. Patients' enrollment will be competed among different sites, but futher step should be taken only after the 3 patients in one group complete the first cycle, their efficacy and safety have been completely evaluated, and the notification of going to next step by a CRO company.

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-sen University Cancer Centre, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang XX, Gao Y, Jin J, Cao JN, Feng JF, Wang HQ, Zhang HL, Cai QQ, Li ZM, Jiang WQ, Huang HQ; Lymphoma Committee, Chinese Anti-Cancer Association (CACA). Bortezomib in combination with fludarabine plus cyclophosphamide for patients with relapsed or refractory mantle-cell lymphoma: results of the LYM-4003 study. Ann Hematol. 2021 Dec;100(12):2961-2968. doi: 10.1007/s00277-021-04619-4. Epub 2021 Jul 31. PMID 34331111